CLINICAL TRIAL: NCT07170176
Title: The Impact of Percutaneous Patent Foramen Ovale Closure on Glymphatic Function and Clinical Symptoms in Patients With Migraine
Brief Title: Effects of PFO Closure on Glymphatic Function and Clinical Symptoms in Patients With Migraine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJTUIAF2025LSYY-609
Record Dates: First submitted 2025-09-07; First posted 2025-09-12 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Migraine Disorders; Patent Foramen Ovale; Right-to-Left Shunt, Cardiac
Keywords: Patent Foramen Ovale; Migraine; Glymphatic System; PFO Closure
MeSH Terms: conditions — Migraine Disorders; Foramen Ovale, Patent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PFO with Migraine (Closure) (Experimental): Patients with patent foramen ovale (PFO) and migraine receive percutaneous PFO closure intervention. This group will be assessed for migraine symptoms and glymphatic function before and after the procedure.
  Interventions: Device: Percutaneous Patent Foramen Ovale Closure
- PFO without Migraine (Observation) (Other): Patients with patent foramen ovale (PFO) but without migraine. This group does not receive closure intervention and serves as the control group for observational comparison. They will undergo the same assessment schedule as the intervention group.
  Interventions: Other: No Intervention

INTERVENTIONS:
Device: Percutaneous Patent Foramen Ovale Closure — Percutaneous transcatheter closure of patent foramen ovale (PFO) is a minimally invasive procedure. Under local anesthesia, a closure device is delivered via a catheter through the femoral vein to the heart to seal the PFO tunnel. The procedure is performed under fluoroscopic and echocardiographic guidance. This intervention aims to eliminate right-to-left shunt, which is hypothesized to improve migraine symptoms and glymphatic function.
  Other Names: PFO Closure
  Arms: PFO with Migraine (Closure)
Other: No Intervention — This arm does not receive the PFO closure procedure. Patients in this control group are observed under their standard care regimen without any study-specific intervention.
  Arms: PFO without Migraine (Observation)

SUMMARY:
Patent Foramen Ovale (PFO) is a common congenital heart defect. Recent studies have suggested a potential association between PFO and migraines, particularly migraine with aura. It is hypothesized that PFO may allow microemboli or vasoactive substances from venous blood to bypass pulmonary metabolism and enter the arterial system directly, potentially triggering migraines. Although PFO closure has been shown to reduce the frequency and severity of migraine attacks, its long-term efficacy and underlying mechanisms require further investigation.

This study aims to explore the characteristics of glymphatic system function in PFO patients and its relationship with migraine symptoms, as well as the impact of PFO closure on glymphatic function and its role in alleviating migraine symptoms. A case-control and self-controlled before-after study design is adopted. Two groups of participants are enrolled: a case group consisting of PFO patients with significant right-to-left shunt and migraine, and a control group comprising PFO patients with significant shunt but without migraine. According to clinical guidelines and after obtaining informed consent, eligible patients in the case group undergo percutaneous PFO closure.

By comparing migraine symptoms and glymphatic function indicators both before and after the procedure between the two groups, the interventional effect of PFO closure and its potential mechanism will be investigated. The primary endpoint is the improvement in migraine symptoms, while the secondary endpoints include glymphatic function metrics. The findings of this study will provide new theoretical insights and clinical guidance for the management of PFO-related migraines.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 to 60 years.
2. Diagnosed with patent foramen ovale (PFO) with significant right-to-left shunt.
3. For the case group: Diagnosis of migraine (with or without aura) according to the International Classification of Headache Disorders (ICHD-3).
4. For the control group: No history of migraine.
5. Willing and able to provide written informed consent.
6. Education level of primary school or higher.

Exclusion Criteria:

1. Patients with a history of PFO closure or other migraine-related surgical treatments;
2. Patients with other severe cardiac or neurological diseases, mental disorders, or psychological conditions;
3. Patients with contraindications to closure surgery or MRI scans (e.g., severe infection, coagulation dysfunction, cardiac pacemakers, aneurysm clips, metallic foreign bodies in the eye, non-removable metal dentures, etc.);
4. Patients unable to complete migraine symptom assessments or imaging examinations due to other reasons.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-14 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Monthly Migraine Days (MMD) | For the intervention arm, this is 6 months post-procedure. For the control arm, this is 6 months post-enrollment.
  The number of days with migraine headache per month, as recorded by participants in a daily headache diary. The change in MMD from baseline to 6-month follow-up will be calculated. A decrease in MMD indicates improvement.

SECONDARY OUTCOMES:
Migraine Pain Intensity (VAS Score) | The pain intensity of migraine attacks as measured by the Visual Analogue Scale (VAS), ranging from 0 (no pain) to 10 (worst pain imaginable). The change in VAS score from baseline to the 6-month timepoint will be calculated. A negative change indicates
  The change in pain intensity of migraine attacks as measured by the Visual Analogue Scale (VAS), ranging from 0 (no pain) to 10 (worst pain imaginable). A negative change indicates improvement.
DTI-ALPS Index | For the intervention arm, this is 6 months post-procedure. For the control arm, this is 6 months post-enrollment.
  The Diffusion Tensor Imaging-Alignment along the Perivascular Space (DTI-ALPS) index is a non-invasive MRI biomarker used to assess glymphatic system function. It is calculated by obtaining diffusion tensor imaging (DTI) sequences on a 3.0T MRI scanner and measuring the diffusion coefficients along the x, y, and z axes in specific regions of interest (ROIs) near the lateral ventricles. The change in the DTI-ALPS index from baseline to the 6-month timepoint will be calculated. A positive change suggests improved glymphatic activity.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Luoyang Central Hospital, Luoyang, Henan
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality